CLINICAL TRIAL: NCT07353606
Title: Determination of Cofilin-2 (rs80358250) and Lactoferrin (rs1126478) Genetic Polymorphism and Change in Their Protein Levels Before and After Non-surgical Periodontal Therapy in Periodontitis Patients With and Without Coronary Heart Disease - An Interventional Study.
Brief Title: Cofilin-2 (rs80358250) and Lactoferrin (rs1126478) Polymorphism and Protein Levels With Non Surgical Periodontal Therapy in Periodontitis Patients With and Without CHD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor and Head, Department of Periodontics, Meenakshi Ammal Dental College and Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MADCH/IEC-II/48/2024
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Periodontitis; Chronic Periodontitis (Disorder); Coronary Heart Disease
Keywords: chronic periodontitis; coronary heart disease; cofillin-2; lactoferrin
MeSH Terms: conditions — Periodontitis; Chronic Periodontitis; Coronary Disease | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP I: 21 systemically healthy subjects with healthy periodontium. (Experimental): Systemically healthy subjects with healthy periodontium having probing pocket depth (PPD) ≤3mm, no clinical attachment loss (CAL=0) and bleeding on probing ≤ 10% of sites.
  Interventions: Procedure: Scaling and root planing
- GROUP II: 21 periodontitis patients without coronary heart disease (Experimental): Systemically healthy subjects with periodontitis having interdental clinical attachment loss ≥ 3-5mm (stage II/III periodontitis) and probing pocket depth (PPD) ≥5mm (stage II/III periodontitis) and bleeding on probing ≥10% of sites.
  Interventions: Procedure: Scaling and root planing
- GROUP III: 21 coronary heart disease patients without periodontitis (Experimental): Patients diagnosed with coronary artery disease with healthy periodontium having probing pocket depth (PPD)≤3mm, no clinical attachment loss (CAL=0) and bleeding on probing ≤ 10% of sites (CAD).
  Interventions: Procedure: Scaling and root planing
- Group IV: 21 periodontitis patients with coronary heart disease. (Experimental): Coronary heart disease (CHD) patients with periodontitis having interdental clinical attachment loss ≥3-5mm (stage II/III periodontitis) and probing pocket depth (PPD) ≥5mm (stage II/III periodontitis) and bleeding on probing ≥ 10%.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Scaling and root planing is a deep cleaning below the gumline used to treat gum disease. Gum disease is caused by a sticky film of bacteria called plaque. Plaque is always forming on your teeth, but if they aren't cleaned well, the bacteria in plaque can cause your gums to become inflammed.

SUMMARY:
Periodontitis is a chronic multifactorial inflammatory disease associated with the accumulation of dental plaque and characterized by progressive destruction of the teeth-supporting apparatus, including the periodontal ligament and alveolar bone. Dental plaque accumulation at the gingival margin initiates an inflammatory response that, in turn, causes microbial alterations and may lead to drastic consequences in the periodontium of susceptible individuals. The pathophysiology of periodontitis is influenced by the relationship between the host immune system and periodontal pathogens. The presence of periodontal pathogens and their metabolic by-products in the oral cavity may get disseminated to the systemic circulation which may pose a risk for various systemic diseases such as cardiovascular disease, oral and colorectal cancer, gastrointestinal diseases, respiratory tract infection, adverse pregnancy outcomes and diabetes.

Although pathogenic bacteria and various other environmental factors are involved in pathogenesis of periodontitis, genetic factors are also known to play a pivotal role in influencing the inflammatory and immune response. Genetic polymorphisms are alterations in the DNA sequence found in general population. Most forms of periodontitis represent a life-long account of interactions between the genome and the environment. The previous literature has stated a strong association of genetic polymorphisms in periodontitis and coronary artery diseases. Identifying these polymorphisms can potentially lead to a better understanding of the mechanisms modulating the expression of inflammatory mediators as well as provides potential therapeutic targets in the prevention of periodontal disease. Two such novel polymorphisms have gained attention recently, namely the Cofilin-2 and Lactoferrin polymorphisms.

Cofilin is one of the most affluent and common actin-binding proteins and plays a role in cell motility, migration, shape, and metabolism. They also play an important role in severing actin filament, nucleating, depolymerizing and bundling activities. Cofilin is the major ADF/cofilin isoform in mammalian neurons influences the dynamics of actin assembly by severing or stabilizing actin filaments. Cofilin-2 is the only isoform present in mature skeletal muscles. It is composed of 5 α helices, 5 β sheets, and 1 C-terminal β short chain, with a molecular weight of 18 kDa. Cofilin-2 is a member of the AC group of proteins that also includes cofilin-1 and destrin, all of which regulate actin-filament dynamics. Recently, Cofilin 2 gained attention as an emerging biomarker for coronary heart diseases. Cofilin-2 has shown to play a role in pathophysiology of coronary heart disease.

Lactoferrin is a multifunctional protein of the transferrin family. Lactoferrin is a globular glycoprotein with a molecular mass of about 80 kDa that is widely represented in various secretory fluids, such as milk, saliva, tears and nasal secretions. Lactoferrin, a multifunctional iron-binding glycoprotein, is involved in coronary heart disease pathophysiology. Recent studies reported that Lactoferrin polymorphism is associated with an increased risk of coronary artery disease in the elderly population.

Studies have been done to identify Lactoferrin genetic polymorphisms, however none of the studies have explored the role of Lactoferrin (rs1126478) and its protein level in subjects with both periodontal disease and coronary heart disease occurring as a continuum. Its expression in periodontitis and coronary heart disease patients is yet to be explored. Genetic polymorphism and protein levels of Cofilin-2 (rs80358250) has been never studied in coronary heart disease and periodontitis. This may further improve our understanding of the influence of this polymorphism on the above mentioned systemic diseases.

NEED FOR THE STUDY While there are studies which have demonstrated the expression of Cofilin-2 and Lactoferrin polymorphisms in various inflammatory conditions, there are no studies to state their expression in the subgingival plaque samples of periodontitis patients with coronary artery disease, specifically before and after non-surgical therapy. Also, the correlation of both these polymorphisms and their levels with periodontal and cardiac parameters has never been investigated so far. It is suggested that these polymorphisms may play a role as putative risk indicators in periodontitis subjects with coronary heart disease which may alter following non-surgical periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient willing to participate in the study.
2. Male and female patients with the age group of 30 to 65 years.
3. Patient having more than or equal to 10 remaining natural teeth.
4. No history of long-term antibiotic use in past 6 months.

Exclusion Criteria:

1. Subjects with systemic conditions such as type I and type II diabetes mellitus, respiratory diseases, renal disease, liver disease, rheumatoid arthritis, allergy, advanced malignancies/neoplasm and HIV infection will be excluded from the present investigation.
2. Subjects on drugs such as corticosteroids or antibiotics within 6 months of investigation or antiepileptic drugs (phenytoin or cyclosporine) having an impact on periodontal tissues will be excluded.
3. Pregnant women (pregnancy may alter the oral flora).
4. Current smokers and individuals who quit smoking less than 6 months.
5. Patients who have undergone periodontal therapy within the previous 6 months.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Changes in periodontal parameters | Baseline-24 months
  Change in periodontal probing depth (measured in mm higher value indicate disease progression)
Change in periodontal variables | Baseline - 2 years
  Change in Clinical attachment level (measured in mm higher value indicate disease progression)
Change in periodontal criteria | Baseline - 2 years
  Change in plaque index (measured as a ratio, range: 0 to 3, maximum value indicates worse outcome and minimum value indicates better outcome)
Change in periodontal variables | Baseline - 2 years
  Changes in Gingival index (measure as a ratio, (0-3)higher value indicates severity of gingival inflammation)

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Kilpauk medical college and hospital, Chennai, Tamil Nadu
  - Meenakshi Ammal Dental College and hospital, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeng Q, Fang Q, Zhou X, Yang H, Dou Y, Zhang W, Gong P, Rong X. Cofilin 2 Acts as an Inflammatory Linker Between Chronic Periodontitis and Alzheimer's Disease in Amyloid Precursor Protein/Presenilin 1 Mice. Front Mol Neurosci. 2021 Sep 30;14:728184. doi: 10.3389/fnmol.2021.728184. eCollection 2021. PMID 34658785
- [Background] Nguyen K, Chau VQ, Mauro AG, Durrant D, Toldo S, Abbate A, Das A, Salloum FN. Hydrogen Sulfide Therapy Suppresses Cofilin-2 and Attenuates Ischemic Heart Failure in a Mouse Model of Myocardial Infarction. J Cardiovasc Pharmacol Ther. 2020 Sep;25(5):472-483. doi: 10.1177/1074248420923542. Epub 2020 May 11. PMID 32390525